CLINICAL TRIAL: NCT03456999
Title: A Randomized, Double Blind, Placebo Controlled Study to Assess the Safety, Tolerability, and Efficacy of MAU868 for the Prevention of Allograft-threatening BK Virus Infection in Kidney Transplant Recipients
Brief Title: Determine the Safety, Tolerability, and Efficacy of MAU868 for the Prevention of BK Virus Infection in Kidney Transplant Recipients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: company decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CMAU868X2201
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: BK Virus Nephropathy
Keywords: BKV, renal transplant, renal and kidney transplant

STUDY DESIGN:
Intervention Model Description: This is a non-confirmatory, randomized, placebo-controlled, blinded, proof-of-concept study in kidney transplant recipients. Approximately 96 eligible patients are planned to be randomized 2:1 to receive MAU868 or placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a patient, investigator and sponsor-blinded study. Patients and investigators will remain blinded to study treatment throughout the study,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MAU868 (Active Comparator): BKV-specific, pan-serotype neutralizing antibody
  Interventions: Biological: MAU868
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MAU868 — MAU868 infused i.v. over 1 hour. One dose will be administered monthly for a total of 6 doses.
  Arms: MAU868
Biological: Placebo — Solution containing no active excipients, infused i.v. over 1 hour. One dose will be administered monthly for a total of 6 doses
  Arms: Placebo

SUMMARY:
This study is being conducted to determine whether MAU868 warrants further clinical development for the prevention of BKV infection in kidney transplant recipients.

DETAILED DESCRIPTION:
This is a non-confirmatory, randomized, placebo-controlled, blinded, proof-of-concept study in kidney transplant recipients. Approximately 96 eligible subjects are planned to be randomized 2:1 to receive MAU868 or placebo. At least 78 subjects are expected to complete the study. The study will consist of a pre-treatment (screening) consenting period, a 24 week treatment period (consisting of 6 monthly i.v. doses of MAU868 or placebo) and a 24 week follow-up period. Subjects who complete the study per protocol will attend a total of 16 visits over a period of 48 weeks.

ELIGIBILITY:
Inclusion criteria;

* Male or female recipients of a first or second kidney or kidney-pancreas transplant who weigh at least 30 kg and are at least 7 years of age (in the US, 18 years of age or above) at the time of transplantation.
* Recipients of organs from a heart-beating deceased, non-heart-beating deceased, living unrelated, or human leukocyte antigen (HLA)-mismatched living related donor.
* Recipients who are treated with lymphocyte-depleting induction therapy (e.g., rabbit antithymocyte globulin, alemtuzumab). Subjects treated with rabbit antithymocyte globulin must receive a total dose of at least 3 mg/kg. Subjects treated with alemtuzumab must receive a total dose of at least 20 mg.
* Recipients of a kidney with a cold ischemia time (CIT) <36 hours.

Exclusion Criteria:

* Recipients of organs from identical twins or living, HLA-matched, related donors.
* ABO incompatible or complement-dependent lymphocytotoxic (CDC) crossmatch positive transplant (isolated positive B cell crossmatches are not an exclusion criterion).
* Recipients who are treated with non-lymphocyte-depleting induction therapy (e.g., basiliximab) or no induction therapy.
* Recipients who are treated or planned to be treated with mTOR inhibitors as part of their initial immunosuppression regimen post-transplantation.
* Recipients who require antibody-depletion prior to transplantation and in the opinion of the investigator are likely to require antibody-depletion after transplantation. Antibody-depleting therapies include but are not necessarily limited to plasmapharesis, immunoadsorption, and IVIg.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by hCG testing.
* Current clinical, radiographic, or laboratory evidence of active or latent tuberculosis (TB) or any history, in the opinion of the investigator, that confers a risk of reactivation of TB and precludes the use of conventional immunosuppression.
* History of splenectomy or asplenia.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using basic methods of contraception during dosing of investigational drug.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2020-07-13 (Estimated); Study Completion 2020-11-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of BK viremia | 24 weeks
  >1000 copies/mL through 24 weeks

SECONDARY OUTCOMES:
Pharmacokinetics of MAU868 | 48 weeks
  Cmin
Immunogenicity of MAU868 | 48 weeks
  Investigate the potential development of anti-drug antibodies